CLINICAL TRIAL: NCT03269019
Title: Thrombotic Biomarkers to Predict Thrombosis in Heparin-induced Thrombocytopenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017CX05
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Heparin-Induced Thrombocytopenia; Thrombosis; Biomarkers
Keywords: Heparin-induced thrombocytopenia; Thrombosis; thrombin-antithrombin; d-dimer; Thrombelastograghy
MeSH Terms: conditions — Thrombosis | interventions — Blood Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIT-group: The patients with heparin-induced thrombocytopenia.
  Interventions: Diagnostic Test: HIT with thrombosis
- HITTs-group: The patients with heparin-induced thrombocytopenia with thrombosis.
  Interventions: Diagnostic Test: HIT with thrombosis
- Control group: The patients without heparin-induced thrombocytopenia and heparin-induced thrombocytopenia with thrombosis.

INTERVENTIONS:
Diagnostic Test: HIT with thrombosis — Testing thrombin-antithrombin complex, d-dimer, fibrin degradation products and Thrombelastograghy.
  Groups: HIT-group; HITTs-group

SUMMARY:
Heparin induced thrombocytopenia (HIT) is a kind of catastrophic thrombotic complications after the application of heparin. If HIT without treatment, death rate is as high as 30% to 50%. Early diagnosis of HIT and prevention of thrombosis is very important.

This study is planned to assess the use of thrombotic biomarkers in patients with HIT, including thrombin-antithrombin complex, d-dimer, fibrin degradation products and Thrombelastograghy monitoring . These biomarkers are monitored in 5-14 days post-operation to assess the risk of thrombosis in HIT patients. All patients were followed up for 30 days, and clinical outcomes, including new thrombus and death, were recorded during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients undergoing cardiac surgery.
* Receiving unfractionated heparin anticoagulation.

Exclusion Criteria:

* history of heparin-induced thrombocytopenia
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are those who receiving cardiac surgery, including valve replacementheart,Coronary Artery Bypass Grafting,aorta replacement etc.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-11-20 (Estimated); Primary Completion 2019-08-19 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Thrombotic event | 30 days
  New thrombosis, including deep venous thrombosis,pulmonary embolism,Cerebral infarction,superior mesenteric artery embolism,artery embolism etc.
Deaths | 30 days
  All-cause deaths

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlu Zhang, MD,Ph.D, Study Director — Wuhan Asia Heart Hospital

IPD SHARING:
Plan to Share IPD: Undecided
We are going to make individual participant data (IPD) available to other researchers after our paper published.